CLINICAL TRIAL: NCT01412697
Title: Fruit and Vegetable Intake Among Rural Youth Following a School-based Randomized Controlled Trial
Brief Title: An Intervention Targeting Fruit and Vegetable Intake Among Rural Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #8520369
Record Dates: First submitted 2011-08-03; First posted 2011-08-09 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Imbalance of Constituents of Food Intake
Keywords: Rural youth; Theory-based intervention; Randomized by schools; Fruit and vegetable intake; Health classes
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fruit and Vegetable Intake Behavioral Intervention (Experimental): measure fruit and vegetable intake in rural youth based on specific behavioral intervention.
  Interventions: Behavioral: Fruit and vegetable intake in rural youth
- Control Group (No Intervention): control group received the standard health information

INTERVENTIONS:
Behavioral: Fruit and vegetable intake in rural youth — A theory based health behavior intervention, developed for youth is presented to seventh grade youth over 8 weeks to test their improvement in their intake of fruits and vegetables.
  Arms: Fruit and Vegetable Intake Behavioral Intervention

SUMMARY:
The investigators implemented a theory-based randomized controlled trial in ten rural Virginia middle schools in 2008-2010 and assessed the impact on health behaviors including fruit/vegetable intake as a primary outcome. Schools were randomized to intervention or control groups. Goal setting, peer leaders, and in-class workshops were intervention features. Seventh graders filled out surveys on health behaviors, psycho-social variables, and demographic characteristics. The investigators expected schools receiving the intervention to report a higher fruit-vegetable intake compared to control schools where students received standard health information. Sample (n=1,119) was 48.5% female, 50% White, with a mean age of 12.6 years. Fruit/vegetable intake was significantly higher in intervention schools at immediate post and at 1-year follow-up compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* 7 grade youth
* attending participating middle schools

Exclusion Criteria:

* In grades other than 7th grade

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1119 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Fruit and vegetable intake | Up to one year
  We surveyed students on fruit/vegetable intake at baseline, immediate post intervention and 1 year follow-up

SECONDARY OUTCOMES:
Confidence to increase fruit and vegetable intake | Up to one year
  We surveyed students on their confidence in increasing their daily servings of fruit and vegetalbes.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Danish, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Nottoway Middle School, Crewe, Virginia, United States

REFERENCES:
- [Derived] Wilson DB, Jones RM, McClish D, Westerberg AL, Danish S. Fruit and vegetable intake among rural youth following a school-based randomized controlled trial. Prev Med. 2012 Feb;54(2):150-6. doi: 10.1016/j.ypmed.2011.11.005. Epub 2011 Dec 3. PMID 22178819